CLINICAL TRIAL: NCT01892397
Title: Pilot Study of Optune (NovoTTF-100A) for Recurrent Atypical and Anaplastic Meningioma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: NovoCure Ltd. (Industry); Columbia University (Other); University of Cincinnati (Other); University of Colorado, Denver (Other); University of Miami (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-067
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Brain Cancer
Keywords: intracranial supratentorial meningioma; Atypical and Anaplastic Meningioma; Optune (NovoTTF-100A); 13-067
MeSH Terms: conditions — Brain Neoplasms; Meningioma

ARMS (1):
- Optune (NovoTTF-100A) (Experimental): The treatment plan is to have patients use the Optune device in monotherapy for ≥ 18 hours per day as per the treatment standard established from prior studies. A medical professional will see each patient at least once per month while on the device for toxicity assessment, compliance evaluation via downloading of the log-file on the device by the Novocure technician (which involves the technician simply attaching the device to a computer via USB where software reads how many hours per day on each day the device was used), and physical examination. Extent of disease evaluations will occur at baseline, 8 weeks, and then every 8 weeks thereafter. These evaluations will include MRI of the brain with and without contrast and perfusion (or CT head if a patient cannot undergo MRI).
  Interventions: Device: Optune (NovoTTF-100A)

INTERVENTIONS:
Device: Optune (NovoTTF-100A)

SUMMARY:
The purpose of this study is to find out what effects, good or bad, the Optune device has on the patient and meningioma. This study is being done because currently there are no proven effective medical treatments for a progressive meningioma that has failed surgery and/or radiation. The study uses an experimental device called Optune. Optune is "experimental" because it has not been approved by the U.S. Food and Drug Administration (FDA) for this type of tumor, although it has been approved for a different type of brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven recurrent WHO grade II (atypical) or grade III (anaplastic) intracranial supratentorial meningioma. MSKCC central review of histology is not required.
* Unequivocal evidence for tumor progression by MRI with and without contrast and with perfusion (or CT scan is MRI with contraindicated). The scan must be performed within 14 days of registration.
* Patients must be on a stable or decreased dose of steroids for at least 5 days prior to baseline imaging
* Patients with recent resection for recurrent disease must have recovered from the effects of surgery and should not start treatment for at least 28 days after surgery.
* Patients must have measurable disease, defined as at least 1cm x 1 cm of contrast enhancing disease.
* Patients must have received prior radiotherapy for meningioma. Patients may have received standard external beam radiation, interstitial brachytherapy, or radiosurgery in any combination. An interval of > 4 weeks (28 days) must have elapsed from the completion of radiotherapy to study entry and there must be subsequent evidence of tumor progression. Patients with prior interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based on PET, MR-perfusion, MR-spectroscopy, or surgical documentation of disease. If there is any question, investigators should discuss with the MSKCC PI.
* Prior therapy: there is no limit on the number of prior surgeries, radiation therapy treatments, radiosurgery treatments, or chemotherapy.
* All patients must be able to provide informed consent indicating that they are aware of the investigational nature of the study. Patients must provide an authorization for the release of their protected health information.
* Age > or = to 18 years old
* Karnofsky performance status > or = to 60%
* 4 weeks (28 days) from any radiation treatment, stereotactic radiosurgery, conventional surgery, or chemotherapy.
* Life expectancy at least 3 months
* Patients with NF (Neurofibromatosis) are eligible, and may have other stable CNS tumors, such as schwannoma, acoustic neuroma, or ependymoma, but ONLY if these lesions have been stable in size for the preceding 6 months.

Exclusion Criteria:

* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix, unless in complete remission and off all therapy for the disease for a minimum of 3 years).
* Concomitant use of any other investigational drugs.
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials (i.e. Quality of life) are allowed.
* Pregnancy or breast feeding. Patients must be surgically sterile, postmenopausal, or agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate. Male patients must be surgically sterile or agree to effective contraception. Female patients of child bearing potential (ages 11-55) must have a negative B-HCG pregnancy test documented within 14 days prior to registration.
* Implanted medical device such as a pacemaker, defibrillator, deep brain stimulator, or vagus nerve stimulator, or documented significant arrhythmia at the discretion of the investigator.
* Evidence of increased intracranial pressure (midline shift >5mm, clinically significant papilledema, vomiting and nausea, or reduced level of consciousness).
* Infratentorial meningioma (patients may have infratentorial meningioma if there is concurrent growing supratentorial meningioma that serves as the target lesion)
* Coagulopathy (as evidenced by PT or APTT >1.5 times upper limit of normal in patients not undergoing anticoagulation)
* Thrombocytopenia (platelet count <100x10^3/uL) Neutropenia (absolute neutrophil count <1x10^3/uL)
* Severe acute infection
* Skull defect with missing bone
* Ventricular shunt/catheter
* Presence of a foreign body intracranially such as a bullet fragment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
progression-free survival rate | 6 months
  From the treatment start date to the date of the first observation of progressive disease (including clinical progression) or death due to any cause. Patients not known to be progression-free at 6 months will be considered treatment failures.

SECONDARY OUTCOMES:
overall survival | 2 year
  From the treatment start date to date of death of any cause.
safety and tolerability | 2 years
  graded according to most up-to-date CTCAE version

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaley, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - University of Miami, Miami, Florida
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/